CLINICAL TRIAL: NCT01194778
Title: Comparison of Efficacy of Different Dosages Vitamin K2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr. C. Vermeer, Maastricht UMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-3-078
Record Dates: First submitted 2010-08-05; First posted 2010-09-03 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-09

CONDITIONS: Carboxylation Level; Vitamin K-dependent Proteins
MeSH Terms: interventions — Vitamin K 1; Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- placebo (Placebo Comparator): The participants of the placebo group will receive daily 1 placebo sachet containing only sucrose
  Interventions: Dietary Supplement: placebo
- vitamin K1 (Active Comparator): The participants of this group will receive daily 1 sachet containing 15 µg vitamin K1.
  Interventions: Dietary Supplement: vitamin K1
- vitamin K2 - 15 µg (Active Comparator): The participants of this group will receive daily 1 sachet containing 15 µg vitamin K2
  Interventions: Dietary Supplement: vitamin K2
- vitamin K2 - 30 µg (Active Comparator): The participants of this group will receive daily 1 sachet containing 30 µg vitamin K2
  Interventions: Dietary Supplement: vitamin K2
- vitamin K2 - 45 µg (Active Comparator): The participants of this group will receive daily 1 sachet containing 45 µg vitamin K2.
  Interventions: Dietary Supplement: vitamin K2

INTERVENTIONS:
Dietary Supplement: placebo — 1 placebo sachet per day containing only sucrose during 12 weeks
  Arms: placebo
Dietary Supplement: vitamin K1 — 15 µg vitamin K1 per day during 12 weeks
  Arms: vitamin K1
Dietary Supplement: vitamin K2 — 15 µg vitamin K2 per day during 12 weeks
  Arms: vitamin K2 - 15 µg
Dietary Supplement: vitamin K2 — 30 µg vitamin K2 per day during 12 weeks
  Arms: vitamin K2 - 30 µg
Dietary Supplement: vitamin K2 — 45 µg vitamin K2 per day during 12 weeks
  Arms: vitamin K2 - 45 µg

SUMMARY:
Vitamin K is a group name for a number of compounds: K1 is present in chloroplasts in green vegetables, K2 is of microbial origin. Lactic bacteria produce a mixture of higher menaquinones, including menaquinone-7, menaquinone-8, and menaquinone-9. Nothing is known yet about the efficacy of bacterial K2 vitamins for in vivo K function (carboxylation of essential proteins). Therefore, this study was undertaken to study effects of different dosages of bacterial vitamin K2 on carboxylation of extrahepatic proteins.

DETAILED DESCRIPTION:
Vitamin K is a group name for a number of compounds: K1 is present in chloroplasts in green vegetables, K2 is of microbial origin. Lactic bacteria produce a mixture of higher menaquinones, including menaquinone-7, menaquinone-8, and menaquinone-9. Higher menaquinones not only have very long half-life times (over 3 days rather than 1 hour for vitamin K1); K2 vitamins are also transported to extra hepatic tissues such as bone and vessel wall whereas K1 is preferentially transported to the liver. Nothing is known yet about the efficacy of bacterial K2 vitamins for in vivo K function (carboxylation of essential proteins). This study describes a dose-response experiment for different dosages of bacterial K2 which are compared with one selected dose of K1 and placebo. The efficacy is concluded from the carboxylation of the bone Gla-protein osteocalcin and of the vascular Gla-protein matrix-Gla protein (MGP).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 40 and 60 years old
* Subjects of normal body weight and height according to BMI < 30
* Subjects of Caucasian race
* Subject has given written consent to take part in the study

Exclusion Criteria:

* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects presenting chronic degenerative and/or inflammatory disease
* Subjects presenting diabetes mellitus
* Abuse of drugs and/or alcohol
* Subjects receiving corticoϊd treatment including inhalators
* Subjects using oral anticoagulants
* Subjects using vitamin K containing multivitamins or vitamin K supplements

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The concentration of the circulating biochemical markers matrix-Gla protein and osteocalcin. Both proteins will be measured in their active form (carboxylated form) and their inactive form (undercarboxylated form). | 12 weeks
  The main purpose of the study is to investigate the efficacy of different dosages bacterial vitamin K2 and vitamin K1 on carboxylation degree of the vitamin K-dependent proteins osteocalcin and matrix-gla protein.

SECONDARY OUTCOMES:
the number or type of bacteria in the stool | 12 weeks
  The second purpose of the study is to monitor whether the increased vitamin K intake will change the composition of the intestinal flora, as measured from the collected stools. Vitamin K, notably K2 is produced by a number of colonic bacteria and our principal is interested to learn whether the intake of extra vitamin K will affect the number or type of bacteria in the stool.

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — VitaK BV Maastricht University
Locations (1):
- VitaK BV Maastricht University, Maastricht, Netherlands